CLINICAL TRIAL: NCT02762838
Title: International Multi-center Comparative Double-blind Randomized Clinical Trial of Efficacy and Safety of BCD-055 (JSC "BIOCAD", Russia) and Remicade® in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Comparative Clinical Trial of Efficacy and Safety of BCD-055 and Remicade® in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-055-3
Record Dates: First submitted 2016-04-04; First posted 2016-05-05 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — BCD-055; Infliximab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-055 (Experimental): Patients in this group will receive BCD-055 in a dose of 3 mg/kg on Week 0, Week 2, Week 6, Week 14, Week 22, Week 30, Week 38, Week 46, Week 54.
  Interventions: Biological: BCD-055; Drug: Methotrexate; Drug: Folic acid
- Remicade® (Active Comparator): Patients in this group will receive Remicade® in a dose of 3 mg/kg on Week 0, Week 2, Week 6, Week 14, Week 22, Week 30, Week 38, Week 46, Week 54.
  Interventions: Biological: Remicade®; Drug: Methotrexate; Drug: Folic acid

INTERVENTIONS:
Biological: BCD-055 — BCD-055 is infliximab biosimilar
  Other Names: infliximab
  Arms: BCD-055
Biological: Remicade®
  Other Names: infliximab
  Arms: Remicade®
Drug: Methotrexate — All patients will receive methotrexate in a dose from 10 to 25 mg per week.
Drug: Folic acid — All patients will receive folic acid in a dose of 5 mg per week.

SUMMARY:
BCD-055-3 is international multi-center comparative double-blind randomized clinical trial of efficacy and safety of BCD-055 (JSC "BIOCAD", Russia) and Remicade® in combination with methotrexate in patients with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Active rheumatoid arthritis according to criteria of American College of Rheumatologists (2010), that was diagnosed at least 6 months prior to screening.
* Active rheumatoid arthritis at screening despite of therapy with methotrexate for 3 last months.
* Use of methotrexate in stable dose for at least 4 weeks before screening (10-25 mg per week).
* History of ineffective treatment with basic antiinflammatory drugs (including methotrexate).

Exclusion Criteria:

* Previous therapy of rheumatoid arthritis with monoclonal antibodies (including anti-tumor necrosis factor drugs)
* Felty's syndrome
* Functional status - class IV according to ACR classification (1991)
* Low activity of rheumatoid arthritis (DAS28-CRP(4) index less than 3.2)
* Patient needs corticosteroids in a dose more than 10 mg (recalculated to prednisolone) before signing informed consent.
* Patients needs equal of less than 10 mg prednisolone but the dose was not stable for last 4 weeks prior to infliximab treatment
* Prior use of disease-modifying antirheumatic drugs including methotrexate, sulfasalazin, chloroquine or hydroxychloroquine for up to 4 weeks before randomization.
* Prior use of alkylating agents for up to 12 months prior to signing informed consent.
* Intraarticular use of corticosteroids for up to 4 weeks before randomization.
* Prior use of live or attenuated vaccines for up to 8 weeks before signing informed consent.
* Diagnosis of tuberculosis.
* Body mass more than 130 kg.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Ratio of patients with ACR20 response after 14 weeks of therapy | Week 14
  Ratio of patients who developed a decrease in American College of Rheumatologists (ACR) score by 20% or more after 14 weeks of therapy with study drug

SECONDARY OUTCOMES:
Ratio of patients with ACR20 response after 30 and 54 weeks of therapy | Week 30, Week 54
  Ratio of patients who developed a decrease in American College of Rheumatologists (ACR) score by 20% or more after 30 and 54 weeks of therapy with study drug
Ratio of patients with ACR50 and 70 response after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients who developed a decrease in American College of Rheumatologists (ACR) score by 50% or more and by 70% or more after 14, 30 and 54 weeks of therapy with study drug
Ratio of patients with low activity of rheumatoid arthritis according to index DAS28-CRP(4) after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with low activity of rheumatoid arthritis according to index Disease Activity Score 28 - C-reactive protein (DAS28-CRP(4), score 2.6-3.2) after 14, 30 and 54 weeks of therapy.
Ratio of patients with low activity of rheumatoid arthritis according to index CDAI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with low activity of rheumatoid arthritis according to Clinical Disease Activity Index (CDAI, score 2.9-10.0) after 14, 30 and 54 weeks of therapy.
Ratio of patients with low activity of rheumatoid arthritis according to index SDAI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with low activity of rheumatoid arthritis according to Simplified Disease Activity Index (SDAI, score 3.4-11.0) after 14, 30 and 54 weeks of therapy.
Ratio of patients with remission of rheumatoid arthritis according to index DAS28 after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with remission of rheumatoid arthritis according to index Disease Activity Score 28 (DAS28, score less than 2.6) after 14, 30 and 54 weeks of therapy.
Ratio of patients with remission of rheumatoid arthritis according to index CDAI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with remission of rheumatoid arthritis according to Clinical Disease Activity Index (CDAI, score 0.0-2.8) after 14, 30 and 54 weeks of therapy.
Ratio of patients with remission of rheumatoid arthritis according to index SDAI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with remission of rheumatoid arthritis according to Simplified Disease Activity Index (SDAI, score 0.0-3.3) after 14, 30 and 54 weeks of therapy.
Ratio of patients with remission of rheumatoid arthritis according to ACR-EULAR criteria after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients with low activity of rheumatoid arthritis according to American College of Rheumatologists (ACR)/ European league Against Rheumatism (EULAR) after 14, 30 and 54 weeks of therapy.
Mean SF-36 score at screening and after 14, 30 and 54 weeks of therapy | Screening, Week 14, Week 30, Week 54
  Mean score of quality of life as assessed by Short Form-36 (SF-36) at screening and after 14, 30 and 54 weeks of therapy.
CRP | Screening, Week 14, Week 30, Week 54
  Dynamics of blood level of C-reactive protein (CRP)
ESR | Screening, Week 14, Week 30, Week 54
  Dynamics of Erythrocyte Sedimentation Rate
Roentgenologic characteristics of abnormal joints after 54 weeks of therapy | Week 54
Frequency of AE/SAE | 54 weeks
Frequency of AE 3-4 grade CTCAE | 54 weeks
Frequency of early withdrawals due to AE/SAE | 54 weeks
Percentage of patients who developed binding and neutralizing antibodies to infliximab | Screening, Week 14, Week 30, Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JSC BIOCAD
Locations (39):
- Belarus (4):
  - Institution of Healthcare "9th Municipal Clinical Hospital", Minsk
  - Institution of Healthcare "First Municipal Clinical Hospital", Minsk
  - Institution of Healthcare "Ordena Trudovogo Krasnogo Znameni Regional Clinical Hospital", Minsk
  - Institution of Healthcare "Clinical Hospital of Vitebsk Region", Vitebsk
- India (6):
  - Shalby Hospital, Ahmedabad
  - Sapthagiri Institute of Medical Sciences and Research Centre, Bangalore
  - S.P Medical College & A.G. of Hospitals, Bīkaner
  - Apollo Gleneagles Hospital, Kolkata
  - Noble Hospital, Pune
  - Ruby Hall Clinic, Pune
- Russia (29):
  - Federal State Budgetary Educational Institution of Higher Education "Altai State Medical University", Barnaul
  - Federal State Autonomous Educational Institution of Higher Professional Education "Belgorod State National Research University", Belgorod
  - State Budgetary Institution of Healthcare "Chelyabinsk Regional Clinical Hospital", Chelyabinsk
  - Regional State Autonomous Institution of Healthcare "Irkutsk Municipal Clinical Hospital No. 1", Irkutsk
  - State Autonomous Institution of Healthcare of Kemerovo Region "S. V. Belayev Kemerovo Regional Clinical Hospital", Kemerovo
  - Budgetary Institution of Khanty-Mansi Autonomous Region - Yugra "Regional Clinical Hospital", Khanty-Mansiysk
  - State Budgetary Institution of Healthcare "Research Institute - S. V. Ochapovskiy Regional Clinical Hospital 1, Krasnodar
  - Budgetary Medical Institution "Kursk Regional Clinical Hospital", Kursk
  - Federal State Budgetary Scientific Institution "V. A. Nasonova Research Institute of Rheumatology", Moscow
  - State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University, Moscow
  - State Budgetary Institution of Moscow "O. M. Filatov Municipal Clinical Hospital 15" of the Moscow Healthcare Department, Moscow
  - Private Institution of Healthcare "Railway Clinical Hospital at Nizhniy Novgorod Station of Russian Railways Open-Joint Stock Company", Nizhny Novgorod
  - State Budgetary Institution of Healthcare of Nizhniy Novgorod Region "N. A. Semashko Nizhniy Novgorod Regional Clinical Hospital", Nizhny Novgorod
  - State Autonomous Healthcare Institution of Novosibirsk Region, Municipal Clinic No 1, Novosibirsk
  - Budgetary Institution of Healthcare of Omsk Region "Regional Clinical Hospital", Omsk
  - State Budgetary Institution of Healthcare of the Republic of Karelia "V. A. Baranov Republican Hospital", Petrozavodsk
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University", Rostov-on-Don
  - Federal State Budgetary Educational Institution of Higher Education "I. I. Mechnikov North-West State Medical University", Saint Petersburg
  - Limited Liability Company Baltic Medicine, Saint Petersburg
  - Limited Liability Company BioEq, Saint Petersburg
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg
  - Private Medical Institution Evromedservis, Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "Clinical Rheumatological Hospital 25", Saint Petersburg
  - State Budgetary Institution of Healthcare "Leningrad Region Clinical Hospital", Saint Petersburg
  - Non-state Healthcare Institution "Road Clinical Hospital at Saratov II Station of Russian Railways Open Joint-Stock Company", Saratov
  - State Institution of Healthcare "Regional Clinical Hospital", Saratov
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University", Tomsk
  - State Budgetary Institution of Healthcare of Tyumen Region "Regional Clinical Hospital No. 1", Tyumen
  - State Institution of Healthcare "Municipal Clinical Emergency Hospital 25", Volgograd

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lila AM, Mazurov VI, Denisov LN, Nesmeyanova OB, Ilivanova EP, Eremeeva AV, Usacheva JV, Dokukina EA, Chernyaeva EV, Ivanov RA. A phase III study of BCD-055 compared with innovator infliximab in patients with active rheumatoid arthritis: 54-week results from the LIRA study. Rheumatol Int. 2019 Sep;39(9):1537-1546. doi: 10.1007/s00296-019-04359-9. Epub 2019 Jul 10. PMID 31292709